CLINICAL TRIAL: NCT02579863
Title: A Phase III Study of Lenalidomide and Low-Dose Dexamethasone With or Without Pembrolizumab (MK3475) in Newly Diagnosed and Treatment Naïve Multiple Myeloma (KEYNOTE 185).
Brief Title: Study of Lenalidomide and Dexamethasone With or Without Pembrolizumab (MK-3475) in Participants With Newly Diagnosed Treatment Naive Multiple Myeloma (MK-3475-185/KEYNOTE-185)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to business reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-185; 2015-002901-12 (EudraCT Number); 163239 (Registry Identifier: JAPIC-CTI); MK-3475-185 (Other: Merck); KEYNOTE-185 (Other: Merck)
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Multiple Myeloma
Keywords: PD1; PD-1; PD-L1; PDL1
MeSH Terms: conditions — Multiple Myeloma | interventions — pembrolizumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Lenalidomide + Dexamethasone (Experimental): Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle PLUS lenalidomide 25 mg orally (PO) on Days 1 to 21 of each 21-day treatment cycle, and dexamethasone 40 mg PO on Days 1, 8, 15 and 22 of each 28-day cycle for up to 18 cycles.
  Interventions: Biological: Pembrolizumab; Drug: Lenalidomide; Drug: Dexamethasone
- Lenalidomide + Dexamethasone (Active Comparator): Participants received lenalidomide 25 mg PO on Days 1 to 21 of each 21-day treatment cycle, and dexamethasone 40 mg PO on Days 1, 8, 15 and 22 of each 28-day cycle for up to 18 cycles.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475
  Arms: Pembrolizumab + Lenalidomide + Dexamethasone
Drug: Lenalidomide — oral capsules
Drug: Dexamethasone — oral tablets

SUMMARY:
The purpose of this study is to compare the efficacy of lenalidomide and low dose dexamethasone with pembrolizumab (MK-3475) to that of lenalidomide and low dose dexamethasone without pembrolizumab in terms of progression-free survival (PFS) in participants with newly diagnosed and treatment-naïve multiple myeloma who are ineligible for autologous stem cell transplant (Auto-SCT). The study's primary hypothesis is that pembrolizumab in dexamethasone prolongs progression free survival (PFS) as assessed by Clinical Adjudication Committee (CAC) blinded central review using International Myeloma Working Group (IMWG) response criteria compared to treatment combination with lenalidomide and low-dose with lenalidomide and low-dose dexamethasone (standard of care, SOC) alone.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of active multiple myeloma and measurable disease.
* Ineligible to receive treatment with auto-SCT due to age (≥65 years old) or any significant coexisting medical condition (cardiac, renal, pulmonary or hepatic dysfunction), likely to have a negative impact on tolerability of auto-SCT. Participants <65 years of age who refuse auto-SCT are not eligible for this study.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Female participants of childbearing potential must have 2 negative urine pregnancy tests (with a sensitivity of at least 25 Milli-international units/milliliter) within 10 to 14 days and within 24 hours prior to receiving study medication.
* Female participants of childbearing potential must agree to use adequate contraception 28 days prior to study start, continuing throughout the study, and for up to 28 days after the last dose of lenalidomide (or 120 days after the last dose of pembrolizumab).
* Male participants of childbearing potential must agree to use adequate contraception from the first dose of study medication, continuing throughout the study, and for up to 28 days after the last dose of lenalidomide (or 120 days after the last dose of pembrolizumab).

Exclusion Criteria:

* Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years.
* Has peripheral neuropathy ≥ Grade 2.
* Has a known additional malignancy that is progressing or requires active treatment within the last 5 years (except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy).
* Has history of non-infectious pneumonitis that required steroids or current pneumonitis
* Has received prior therapy with an anti-programmed cell death 1 receptor (anti-PD-1), anti-programmed death-ligand 1 (anti-PD-L1), anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has a known Human Immunodeficiency Virus (HIV), or a known, active Hepatitis B (HBV), or a known, active Hepatitis C (HCV) infection.
* Is unable or unwilling to undergo thromboembolic prophylaxis including, as clinically indicated, aspirin, Coumadin (warfarin) or low-molecular weight heparin.
* Has lactose intolerance.
* Has an invasive fungal infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Usmani SZ, Schjesvold F, Oriol A, Karlin L, Cavo M, Rifkin RM, Yimer HA, LeBlanc R, Takezako N, McCroskey RD, Lim ABM, Suzuki K, Kosugi H, Grigoriadis G, Avivi I, Facon T, Jagannath S, Lonial S, Ghori RU, Farooqui MZH, Marinello P, San-Miguel J; KEYNOTE-185 Investigators. Pembrolizumab plus lenalidomide and dexamethasone for patients with treatment-naive multiple myeloma (KEYNOTE-185): a randomised, open-label, phase 3 trial. Lancet Haematol. 2019 Sep;6(9):e448-e458. doi: 10.1016/S2352-3026(19)30109-7. Epub 2019 Jul 18. PMID 31327689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 140 centers in 15 countries. The database cutoff date was August 3, 2020.
Pre-assignment Details: Note: Due to administrative reasons (a noncompliant site), 2 participants in the Pembrolizumab plus SOC arm and one participant in the SOC arm, were recorded as "Ongoing in Trial" in the CSR Disposition Table and "Final Disposition Unknown" here.
Groups:
- Lenolidomide + Dexamethasone: Participants received lenalidomide 25 mg PO on Days 1 to 21 of each 21-day treatment cycle, and dexamethasone 40 mg PO on Days 1, 8, 15 and 22 of each 28-day cycle for up to 18 cycles.
Period: Overall Study
Arm/Group | Pembrolizumab + Lenalidomide + Dexamethasone | Lenolidomide + Dexamethasone
Started | 156 | 154
Treated | 154 | 148
Completed | 0 | 0
Not Completed | 156 | 154
Not completed — Final Disposition Unknown | 2 | 1
Not completed — Adverse Event | 18 | 11
Not completed — Death | 31 | 29
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Screen Failure | 0 | 2
Not completed — Study Terminated at Selected Sites | 82 | 88
Not completed — Withdrawal by Subject | 20 | 20

BASELINE CHARACTERISTICS:
Population: The analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Lenalidomide + Dexamethasone | Lenolidomide + Dexamethasone | Total
Number analyzed (Participants) | 156 | 154 | 310
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.4 (6.0) | 74.3 (5.9) | 74.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 81 | 166
  Male | 71 | 73 | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 143 | 136 | 279
  Unknown or Not Reported | 9 | 14 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 27 | 54
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 3 | 12
  White | 115 | 121 | 236
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 3 | 6
International Stage (I, II, III). [Number; unit: Participants] — The International Staging System (ISS) defines the factors that influence patient survival. The system has 3 stages based on the measurement of serum albumin and the levels of serum β2-microglobulin (β2-M).
  Stage I: β2-M <3.5 mg/L with a serum albumin of 3.5 g/dL or more;
  Stage II: Either of these 2 criteria:
  β2-M between 3.5 mg/L and 5.5 mg/dL Albumin <3.5 g/dL; Stage III: β2-M >5.5 mg/L.
  Participants
    Stage I | 39 | 53 | 92
    Stage II | 70 | 66 | 136
    Stage III | 46 | 34 | 80
    Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Evaluated According to the International Myeloma Working Group (IMWG) Response Criteria 2011 by Clinical Adjudication Committee (CAC) Blinded Central Review
Description: PFS was defined as the time from randomization to the first documented disease progression (events of new bone lesions, soft tissue plasmacytomas or an increase in existing lesions, or death due to any cause). The median PFS was calculated from the product-limit (Kaplan-Meier) method for censored data. Due to the small number of events, the tail of the estimated survival distribution was close to the median for both arms. The higher variability of the tail estimates resulted in observing the median estimate in the experimental arm but not in the standard of care arm even when number of events in 2 arms were similar. The database cutoff date was July 9, 2018.
Time Frame: Up to approximately 30 months
Population: The analysis population included all randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenalidomide + Dexamethasone | Lenolidomide + Dexamethasone
Number analyzed (Participants) | 156 | 154
Months | 19.6 [15.3 to NA] — Upper Limit could not be estimated due to an insufficient number of events by the date of data cutoff. | NA [15.5 to NA] — The Median was not reached, and the Upper Limit could not be estimated due to insufficient number of events by the date of data cutoff.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenalidomide + Dexamethasone vs Lenolidomide + Dexamethasone; Test type: Superiority; p = 0.33475, Log Rank; One-sided p-value based on Stratified log-rank test; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.56 to 1.45] — Based on Cox regression model with treatment as a covariate stratified by Age (<75 years vs >= 75 years) and ISS stage (I or II vs. III)

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. OS was calculated from the product-limit (Kaplan-Meier) method for censored data. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. This is an event-driven (events of death) outcome measure. At the time of data cut-off, there were an insufficient number of events from the censored data to be able to estimate certain parameters (e.g. medians). The database cutoff date was August 3, 2020.
Time Frame: Up to approximately 55 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenalidomide + Dexamethasone | Lenolidomide + Dexamethasone
Number analyzed (Participants) | 156 | 154
Months | NA [44.6 to NA] — The Median was not reached, and the Upper Limit could not be estimated due to insufficient number of events before the date of data cutoff. | NA [NA to NA] — The Median was not reached, and the Upper and Lower Limits could not be estimated due to insufficient number of events before the date of data cutoff.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenalidomide + Dexamethasone vs Lenolidomide + Dexamethasone; Test type: Superiority; p = 0.83416, Stratified log-rank test; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.81 to 1.84] — Based on Cox regression model with treatment as a covariate stratified by "Age" (<75 years vs >= 75 years) and "ISS stage" (I or II vs. III)

3. Secondary Outcome: Overall Response Rate (ORR) Evaluated According to the IMWG Response Criteria by CAC Blinded Central Review
Description: ORR was based on participants who achieved at least a partial response (stringent complete response [sCR]+complete response [CR]+very good partial response [VGPR]+partial response [PR]) according to the IMWG. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=stringent complete response, CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 hr; PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. The data cutoff date was July 9, 2018.
Time Frame: Up to approximately 30 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Lenalidomide + Dexamethasone | Lenolidomide + Dexamethasone
Number analyzed (Participants) | 156 | 154
Percentage of participants | 74.4 [66.8 to 81.0] | 68.8 [60.9 to 76.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenalidomide + Dexamethasone vs Lenolidomide + Dexamethasone; Test type: Superiority; p = 0.13102, One-sided p-value for testing; H0: difference in % =0 versus H1: difference in % > 0; Difference in % vs SOC = 5.8, 95% CI 2-sided [-4.3 to 15.8]; Based on Miettinen & Nurminen method stratified by 'Age' (<75 years vs >= 75 years) and 'ISS stage' (I or II vs. III); If there were no participants in one of the treatment groups involved in a comparison for a particular stratum, then that stratum was excluded from the treatment comparison

4. Secondary Outcome: Duration of Response (DOR) Evaluated According to IMWG Response Criteria by CAC Blinded Central Review
Description: Response duration was defined as the time from first documented evidence of at least a partial response (sCR+CR+VGPR+PR]), until confirmed disease progression or death. DOR was calculated from product-limit (Kaplan-Meier) method for censored data. This is an event-driven (events of disease progression and death) outcome measure. At the time of data cut-off, there were an insufficient number of events from the censored data to be able to estimate certain parameters (e.g. medians). Full Range is the minimum and maximum of the observed duration of response. The data cutoff date was July 9, 2018.
Time Frame: Up to approximately 30 months
Population: The analysis population included all randomized participants who demonstrated at least a partial response. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenalidomide + Dexamethasone | Lenolidomide + Dexamethasone
Number analyzed (Participants) | 116 | 106
Months | NA [NA to NA] — The Median was not reached, and the limits could not be estimated due to the lack of progressive disease by the time of last disease assessment. | NA [NA to NA] — The Median was not reached, and the limits could not be estimated due to the lack of progressive disease by the time of last disease assessment.

5. Secondary Outcome: Disease Control Rate (DCR) Evaluated According to the IMWG Response Criteria by CAC Blinded Central Review
Description: Disease control rate was defined as the percentage of participants who achieved confirmed sCR, CR, VGPR, PR, or have demonstrated SD for at least 12 weeks prior to any evidence of progression. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 hr; PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours; SD = not meeting the criteria for CR, VGPR, PR, or PD; PD = development of new bone lesions or soft tissue plasmacytomas or on a definite increase in the size of existing bone lesions or soft tissue plasmacytomas. Data cutoff date was July 9, 2018.
Time Frame: Up to approximately 30 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Lenalidomide + Dexamethasone | Lenolidomide + Dexamethasone
Number analyzed (Participants) | 156 | 154
Percentage of participants | 89.1 [83.1 to 93.5] | 91.6 [86.0 to 95.4]

6. Secondary Outcome: Second Progression Free Survival (PFS2)
Description: PFS2 was defined as the time from randomization to subsequent disease progression after initiation of new anti-cancer therapy, or death from any cause, whichever occurred first, by investigator assessment. PFS was assessed by Clinical Adjudication Committee (CAC) blinded central review according to the IMWG response criteria based on the development of new bone lesions or soft tissue plasmacytomas or on a definite increase in the size of existing bone lesions or soft tissue plasmacytomas. PFS2 was not completed due to incomplete enrollment for a clinical hold and study cancellation.
Time Frame: Up to approximately 55 months
Population: The analysis population included all randomized participants. Participants were included in the treatment group to which they were randomized. PFS2 was not completed due to incomplete enrollment for a clinical hold and study cancellation.
Arm/Group | Pembrolizumab + Lenalidomide + Dexamethasone | Lenolidomide + Dexamethasone
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study. The database cutoff date was August 3, 2020.
Time Frame: Up to approximately 55 months
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenalidomide + Dexamethasone | Lenolidomide + Dexamethasone
Number analyzed (Participants) | 154 | 148
Participants | 152 | 141

8. Secondary Outcome: Number of Participants Discontinuing Study Treatment Due to an AE
Description: as for outcome 7
Time Frame: Up to approximately 55 months
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenalidomide + Dexamethasone | Lenolidomide + Dexamethasone
Number analyzed (Participants) | 154 | 148
Participants | 44 | 26

ADVERSE EVENTS:
Time Frame: Up to approximately 55 months
Description: The All-Cause Mortality analysis used all randomized participants whereas adverse events were collected for all treated participants. Disease progression of cancer under study was not considered an adverse event (AE) unless related to study treatment. Medical Dictionary for Regulatory Activities (MedDRA) preferred terms Neoplasm progression, Malignant neoplasm progression and Disease progression not related to study treatment were excluded as AEs. The Database Cutoff Date was Aug. 3, 2020.
Arm/Group | Pembrolizumab + Lenalidomide + Dexamethasone | Lenolidomide + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 51/156 | 43/154
Serious Adverse Events (participants affected / at risk) | 91/154 | 65/148
Other Adverse Events (participants affected / at risk) | 143/154 | 129/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenalidomide + Dexamethasone (N=154) | Lenolidomide + Dexamethasone (N=148)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Cytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0)
Fanconi syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ischaemic enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 3 (3)
Death (General disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 8 (9) | 1 (1)
Sudden death (General disorders) | 1 (1) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (4) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 16 (19) | 10 (10)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 8 (8) | 4 (4)
Septic shock (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 3 (3) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenalidomide + Dexamethasone (N=154) | Lenolidomide + Dexamethasone (N=148)
Anaemia (Blood and lymphatic system disorders) | 32 (48) | 27 (40)
Neutropenia (Blood and lymphatic system disorders) | 30 (54) | 26 (51)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (16) | 12 (19)
Hypothyroidism (Endocrine disorders) | 13 (13) | 1 (1)
Vision blurred (Eye disorders) | 11 (12) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 13 (16) | 13 (18)
Constipation (Gastrointestinal disorders) | 55 (62) | 33 (35)
Diarrhoea (Gastrointestinal disorders) | 36 (51) | 34 (48)
Dry mouth (Gastrointestinal disorders) | 12 (13) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 8 (9) | 2 (2)
Nausea (Gastrointestinal disorders) | 37 (54) | 33 (38)
Stomatitis (Gastrointestinal disorders) | 9 (11) | 6 (6)
Vomiting (Gastrointestinal disorders) | 30 (39) | 9 (16)
Asthenia (General disorders) | 11 (11) | 17 (20)
Fatigue (General disorders) | 44 (52) | 37 (39)
Oedema (General disorders) | 8 (8) | 6 (7)
Oedema peripheral (General disorders) | 25 (31) | 27 (28)
Pyrexia (General disorders) | 29 (41) | 10 (11)
Bronchitis (Infections and infestations) | 9 (12) | 4 (5)
Nasopharyngitis (Infections and infestations) | 11 (16) | 11 (13)
Oral candidiasis (Infections and infestations) | 15 (16) | 2 (2)
Pneumonia (Infections and infestations) | 11 (11) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 13 (17)
Urinary tract infection (Infections and infestations) | 15 (16) | 12 (16)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 8 (10)
Fall (Injury, poisoning and procedural complications) | 7 (10) | 9 (12)
Alanine aminotransferase increased (Investigations) | 11 (11) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 8 (8) | 1 (1)
Neutrophil count decreased (Investigations) | 13 (23) | 12 (23)
Weight decreased (Investigations) | 10 (10) | 17 (18)
Decreased appetite (Metabolism and nutrition disorders) | 26 (28) | 19 (21)
Dehydration (Metabolism and nutrition disorders) | 8 (14) | 5 (6)
Gout (Metabolism and nutrition disorders) | 8 (14) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (17) | 8 (12)
Hypocalcaemia (Metabolism and nutrition disorders) | 16 (18) | 8 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 26 (31) | 17 (21)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (10) | 5 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (10) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (21) | 9 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (24) | 17 (21)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 (17) | 14 (16)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 (12) | 4 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (14) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (11) | 8 (10)
Dizziness (Nervous system disorders) | 14 (15) | 14 (15)
Dysgeusia (Nervous system disorders) | 8 (8) | 12 (12)
Headache (Nervous system disorders) | 9 (9) | 11 (14)
Neuropathy peripheral (Nervous system disorders) | 9 (11) | 12 (13)
Tremor (Nervous system disorders) | 11 (11) | 16 (16)
Anxiety (Psychiatric disorders) | 12 (14) | 11 (12)
Depression (Psychiatric disorders) | 9 (10) | 8 (8)
Insomnia (Psychiatric disorders) | 22 (25) | 27 (33)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 18 (19)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 10 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 12 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (9) | 3 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 8 (10) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (17) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 32 (45) | 19 (20)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 (19) | 11 (13)
Hypotension (Vascular disorders) | 12 (13) | 8 (9)

LIMITATIONS AND CAVEATS:
The MK-3475-185 study was stopped/terminated early. Endpoint statistics may be biased due to the incomplete treatment and follow-up of participants after study termination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT02579863/Prot_SAP_001.pdf